CLINICAL TRIAL: NCT05942027
Title: Clinical Study Evaluating the Role of Coenzyme Q10 as Adjuvant Therapy to Angiotensin Converting Enzyme Inhibitor on Blood Pressure, Proteinuria and Bone Metabolism in Patients With Chronic Kidney Disease
Brief Title: Role of Coenzyme Q10 in Chronic Kidney Disease
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Dina Zaki Mohamed Zaki Abdel Hamid, Clinical Pharmacist, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Coenzyme Q10 in CKD
Record Dates: First submitted 2023-06-26; First posted 2023-07-12 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Chronic Kidney Diseases
Keywords: Proteinuria, Bone Metabolism, Coenzyme Q10
MeSH Terms: conditions — Renal Insufficiency, Chronic; Proteinuria | interventions — coenzyme Q10

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1: Control group (Placebo Comparator): Non-dialysis chronic kidney disease (CKD) patients (Stages 2-3b). Patients will be treated with ramipril 10 mg/day and a placebo match Coenzyme Q10 capsules once per day.The dose of ramipril may be modified according to blood pressure control.
  Participants will be followed-up by weekly telephone calls and monthly direct meetings to assess their adherence for 6 months.
  Interventions: Drug: Placebo
- Group 2: Coenzyme Q10 (Active Comparator): Non-dialysis chronic kidney disease (CKD) patients (Stages 2-3b).Patients will be treated with ramipril 10 mg/day and Coenzyme Q10 capsules (CoQ10) 200 mg/day.The dose of ramipril may be modified according to blood pressure control.
  Participants will be followed-up by weekly telephone calls and monthly direct meetings to assess their adherence for 6 months.
  Interventions: Drug: Co-Enzyme Q10

INTERVENTIONS:
Drug: Placebo — Placebo match Coenzyme Q10 capsules once per day .
  Arms: Group 1: Control group
Drug: Co-Enzyme Q10 — Patients will be treated with Coenzyme Q10 capsules (CoQ10) 200 mg/day.
  Arms: Group 2: Coenzyme Q10

SUMMARY:
This randomized placebo controlled double blind parallel clinical study will be conducted on 44 non-dialysis chronic kidney disease (CKD) patients (Stages 2-3b).Clinical Study Evaluating the Role of Coenzyme Q10 as Adjuvant Therapy to Angiotensin Converting Enzyme Inhibitor on Blood Pressure, Proteinuria and Bone Metabolism in Patients with Chronic Kidney Disease. Patients will be recruited from, Internal Medicine Department, Nephrology Unit, Alexandria Main University Hospital, Egypt. Patients with albumin-to-creatinine ratio ≥ 30 mg/g, with serum Potassium < 5 mEq/L and newly diagnosed patients with hypertension. The study duration will be 6 months. The patients will be randomized using stratified random block method into two groups.

Group 1: Control group Non-dialysis chronic kidney disease (CKD) patients (Stages 2-3b). Patients will be treated with ramipril 10 mg/day and a placebo match Coenzyme Q10 capsules once per day.The dose of ramipril may be modified according to blood pressure control.

Group 2: Coenzyme Q10 Non-dialysis chronic kidney disease (CKD) patients (Stages 2-3b).Patients will be treated with ramipril 10 mg/day and Coenzyme Q10 capsules (CoQ10) 200 mg/day. The dose of ramipril may be modified according to blood pressure control.

Participants will be followed-up by weekly telephone calls and monthly direct meetings to assess their adherence for 6 months.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is defined by a reduction in the kidney function (shown by reduced estimated glomerular filtration rate (eGFR) or markers of kidney damage, or both, for at least three months). It varies depending on the amount of blood pressure control, the degree of proteinuria, the previous rate of decline in GFR, and the underlying renal disease, including diabetes.

Phosphorus excretion decreases in many kidney disorders, and as a result, the amount of fibroblast growth factor 23 (FGF-23) rises.FGF-23 levels have appeared to predict risk of death in individuals with chronic renal disease as the estimated glomerular filtration rate declines, and a corresponding increase in FGF-23 can be noted.

FGF-23 is a hormone with a molecular weight of 30 kDa works on fibroblast growth factor receptors (FGFR1-4) in the kidney, heart, colon, and parathyroid gland. It is secreted by osteocytes and, to a lesser extent by osteoblasts into the bloodstream. A rise in FGF-23 could indicate kidney dysfunction, and concurrent bone disease. Patients with CKD are well known to have greater risk for developing bone fractures.

The term "chronic kidney disease-mineral bone disorder" (CKD-MBD) refers to the decline in bone quality and the subsequent development of disorders in bone and mineral metabolism caused by impaired kidney function. In addition to PTH, vitamin D, calcium and phosphorus, fibroblast growth factor-23 (FGF-23) play a role in CKD-MBD.

Treatment of the underlying disease, if possible, and treatment of secondary factors, such as increased blood pressure and proteinuria, are the two main ways to limit the rate of CKD progression. Angiotensin-converting enzyme (ACE) inhibitors and angiotensin II receptor blockers (ARBs) are renin-angiotensin system (RAS) inhibitors that are more effective than other antihypertensive medications in reducing proteinuria and slowing the rate of progression of proteinuria during CKD, regardless of the etiology.

Ramipril inhibits ACE, which lowers FGF-23 expression in the kidney and attenuates proteinuria. Angiotensin inhibition frequently causes mild to moderate decrease in GFR and hyperkalemia following the treatment initiation or following dose escalation. If CKD is progressive, hyperkalemia may develop quickly after the start of treatment or at a later time.

Coenzyme Q10 (CoQ10) is an organic molecule can be found in both reduced (ubiquinol) and oxidised (ubiquinone) forms in mitochondria and cell membranes. Patients with CKD have been found to have considerably reduced plasma CoQ10 levels. CoQ10 lowers the level of aldosterone and modifies the angiotensin effect on sodium retention. An increase in CoQ10 availability may have altered renin-angiotensin-aldosterone action resulting in a decrease in ACE level. Additionally, the endothelium appears to be directly affected by CoQ10, causing vasodilation and reducing blood pressure. High dose CoQ10 supplementation in cases where the condition is treated early resulted in an improvement in renal function and a reduction in proteinuria.CoQ10 prevent an increase of FGF-23 and also provides a reduction in cardiovascular risk.The aim of this work is to evaluate the role of Coenzyme Q10 (CoQ10) as adjuvant therapy to angiotensin converting enzyme inhibitor on blood pressure, proteinuria and bone metabolism in patients with chronic kidney disease (CKD).

All the participants will be subjected to the following:

1. Demography, History and Physical Examination

* Age, sex, sex distribution ratio (M/F) will be determined. Measurement of weight in nearest kilogram and height in nearest centimeter will be measured using Detecto Scale with subsequent calculation of body mass index according to the following formula: BMI= [Weight (kg) ÷ Height2 (m)]. Full medical history will be taken to avoid inclusion of any patient with confounding disease or medication in the study.
* Measurement of blood pressure will be done using a mercury sphygmomanometer in accordance with recommendations of the American Heart Association and standardized office blood pressure measurements. The mean values of the duplicate measurements will be recorded. The blood pressure will be assessed at baseline and every 4 weeks. Measurements of routine parameters at baseline, through evaluation of:
* Fasting blood glucose
* Alanine aminotransferase (ALT)
* Serum total bilirubin
* In addition, prothrombin time or international normalization ratio (INR) will be also assessed. Assessment of Proteinuria at the time of enrollment, 3 and 6 months after intervention. Proteinuria will be assessed using urine dipstick test. Albumin-to-creatinine ratio will be calculated by dividing the urinary albumin concentration by the urinary creatinine concentration. Assessment of kidney functions at baseline, 4 weeks, 3 and 6 months after initiation of ACEI by assessment: Serum creatinine, Estimated glomerular filtration rate (eGFR) in mL/min/1.73m2 which will be calculated using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) creatinine equation, 2021, blood urea nitrogen and serum potassium Evaluation of Chronic Kidney Disease-Mineral and Bone Disorder Chronic Kidney Disease-Mineral and Bone Disorder (CKD MBD) will be assessed at baseline and at the end of intervention through evaluation of: - Serum level of Fibroblast growth factor-23 (FGF-23)
* Serum Parathyroid hormone (PTH) level .
* Serum concentration of 25 (OH) vitamin D.
* Serum calcium
* Serum phosphorus

Clinical outcome will be assessed at baseline and 6 months after Intervention through:

- Evaluation of Health Related Quality of Life (HRQOL) using the validated Arabic version of -Kidney Disease and Quality of Life- Short Form (KDQOL-SF™) version 1.3 questionnaire which was formerly used in Egypt for patients with CKD.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old.
* Both sexes.
* Patients matched in the duration of CKD.
* Non-dialysis chronic kidney disease (CKD) patient with estimated glomerular filtration rate (GFR) 30-89 mL/min/1.73m2 (Stage 2-3b).
* Patients with albumin-to-creatinine ratio ≥ 30 mg/g.
* Patients with serum Potassium < 5 mEq/L.
* A newly diagnosed patients with hypertension.

Exclusion criteria:

* Patients with elevated level of potassium ≥ 5 mEq/L.
* Patients with diabetes.
* Patients with cancer.
* Patients with heart disease.
* Patients with hepato-biliary disease and other liver diseases.
* Patients with kidney stones and urinary tract infection.
* Patients with an overactive thyroid gland.
* Patients with bleeding disorder.
* History of drug allergy to ACEI or ARBs.
* Pregnant and breastfeeding women.
* Patients with blood pressure ≥180/110 or <100/60.
* Patients on alteplase, azothiopurine, everolimus, sirolimus, lithium, non-steroidal anti-inflammatory drugs (epifenac, tenoxicam, Celecoxib….), potassium retentive diuretics (amiloride, spironolactone), other ACEIs and ARBs will be excluded to avoid possible drug-drug interactions with ramipril.
* Patients on omega-3 fatty acids; vitamins (especially A, C, E, K), Chemotherapy and oral anticoagulant (warfarin), cholestyramine, orlistate will be excluded to avoid possible drug interactions that could affect Coenzyme Q10

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2023-07-15 (Actual); Primary Completion 2026-07-14 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
The change in kidney function test measured by creatinine clearance (eGFR) mL/min/1.73m2 which will be calculated using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) creatinine equation, 2021 | The study duration will be 6 months.
  Assessment of kidney functions at baseline, 4 weeks, 3 and 6 months after initiation of ACEI by assessment: Estimated glomerular filtration rate (eGFR) in mL/min/1.73m2 which will be calculated using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) creatinine equation, 2021.
The change in proteinuria level be assessed using Albumin-to-creatinine ratio (ACR) ratio (mg/g) | The study duration will be 6 months
  Assessment of Proteinuria at the time of enrollment, 3 and 6 months after intervention. Albumin-to-creatinine ratio will be calculated by dividing the urinary albumin concentration by the urinary creatinine concentration (mg/g)
The change in blood pressure (mmHg) will be done using a mercury sphygmomanometer | The study duration will be 6 months
  Measurement of blood pressure will be done using a mercury sphygmomanometer in accordance with recommendations of the American Heart Association and standardized office blood pressure measurements. The mean values of the duplicate measurements will be recorded. The blood pressure will be assessed at baseline and every 4 weeks.
The change in Blood urea nitrogen (BUN) (mg/dl) | The study duration will be 6 months
  Assessment of BUN (mg/dl) at baseline, 4 weeks, 3 and 6 months after initiation of ACEI
The change in serum potassium (meq/l). | The study duration will be 6 months
  Assessment of serum potassium (meq/l) at baseline, 4 weeks, 3 and 6 months after initiation of ACEI
The change in serum creatinine (mg/dl) | The study duration will be 6 months
  Assessment of serum creatinine (mg/dl) at baseline, 4 weeks, 3 and 6 months after initiation of ACEI
The change in serum urea (mg/dl) | The study duration will be 6 months
  Assessment of serum urea (mg/dl) at baseline, 4 weeks, 3 and 6 months after initiation of ACEI

SECONDARY OUTCOMES:
The change in chronic kidney disease-mineral and bone disorder related parameters by assessment Serum level of Fibroblast growth factor-23 (FGF-23) (pg/ml) | The study duration will be 6 months.
  Evaluation of Chronic Kidney Disease-Mineral and Bone Disorder Chronic Kidney Disease-Mineral and Bone Disorder (CKD MBD) will be assessed at baseline and at the end of intervention through evaluation of: - Serum level of Fibroblast growth factor-23 (FGF-23) (pg/ml)
The change in I-PTH (pg/ml) | The study duration will be 6 months
  The change in I-PTH (pg/ml) will be assessed at baseline and at the end of intervention through evaluation
The change in vitamin D level (ng/ml) | The study duration will be 6 months
  The change in vitamin D level (ng/ml) will be assessed at baseline and at the end of intervention through evaluation
The change in serum calcium level (mg/dl) | The study duration will be 6 months
  The change in serum calcium level (mg/dl) will be assessed at baseline and at the end of intervention through evaluation
The change in serum phosphorus level (mg/dl) | The study duration will be 6 months.
  The change in serum phosphorus level (mg/dl) will be assessed at baseline and at the end of intervention through evaluation
Clinical outcome will be assessed by Kidney Disease and Quality of Life- Short Form (KDQOL-SF™) version 1.3 questionnaire | The study duration will be 6 months
  Clinical outcome will be assessed at baseline and 6 months after Intervention through:
  - Evaluation of Health Related Quality of Life (HRQOL) using the validated Arabic version of -Kidney Disease and Quality of Life- Short Form (KDQOL-SF™) version 1.3 questionnaire which was formerly used in Egypt for patients with CKD.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Pharmacy Tanta University, Tanta, Capital of Gharbia Governorate., Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] GBD Chronic Kidney Disease Collaboration. Global, regional, and national burden of chronic kidney disease, 1990-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet. 2020 Feb 29;395(10225):709-733. doi: 10.1016/S0140-6736(20)30045-3. Epub 2020 Feb 13. PMID 32061315
- [Background] Levey AS, de Jong PE, Coresh J, El Nahas M, Astor BC, Matsushita K, Gansevoort RT, Kasiske BL, Eckardt KU. The definition, classification, and prognosis of chronic kidney disease: a KDIGO Controversies Conference report. Kidney Int. 2011 Jul;80(1):17-28. doi: 10.1038/ki.2010.483. Epub 2010 Dec 8. PMID 21150873
- [Background] Isakova T, Xie H, Yang W, Xie D, Anderson AH, Scialla J, Wahl P, Gutierrez OM, Steigerwalt S, He J, Schwartz S, Lo J, Ojo A, Sondheimer J, Hsu CY, Lash J, Leonard M, Kusek JW, Feldman HI, Wolf M; Chronic Renal Insufficiency Cohort (CRIC) Study Group. Fibroblast growth factor 23 and risks of mortality and end-stage renal disease in patients with chronic kidney disease. JAMA. 2011 Jun 15;305(23):2432-9. doi: 10.1001/jama.2011.826. PMID 21673295
- [Background] Shimada T, Hasegawa H, Yamazaki Y, Muto T, Hino R, Takeuchi Y, Fujita T, Nakahara K, Fukumoto S, Yamashita T. FGF-23 is a potent regulator of vitamin D metabolism and phosphate homeostasis. J Bone Miner Res. 2004 Mar;19(3):429-35. doi: 10.1359/JBMR.0301264. Epub 2003 Dec 29. PMID 15040831
- [Background] Sarafidis PA, Khosla N, Bakris GL. Antihypertensive therapy in the presence of proteinuria. Am J Kidney Dis. 2007 Jan;49(1):12-26. doi: 10.1053/j.ajkd.2006.10.014. PMID 17185142
- [Background] Yeung CK, Billings FT 4th, Claessens AJ, Roshanravan B, Linke L, Sundell MB, Ahmad S, Shao B, Shen DD, Ikizler TA, Himmelfarb J. Coenzyme Q10 dose-escalation study in hemodialysis patients: safety, tolerability, and effect on oxidative stress. BMC Nephrol. 2015 Nov 3;16:183. doi: 10.1186/s12882-015-0178-2. PMID 26531095
- [Background] FABRE LF Jr, BANKS RC, MCISAAC WM, FARRELL G. EFFECTS OF UBIQUINONE AND RELATED SUBSTANCES ON SECRETION OF ALDOSTERONE AND CORTISOL. Am J Physiol. 1965 Jun;208:1275-80. doi: 10.1152/ajplegacy.1965.208.6.1275. No abstract available. PMID 14301392
- [Background] Heeringa SF, Chernin G, Chaki M, Zhou W, Sloan AJ, Ji Z, Xie LX, Salviati L, Hurd TW, Vega-Warner V, Killen PD, Raphael Y, Ashraf S, Ovunc B, Schoeb DS, McLaughlin HM, Airik R, Vlangos CN, Gbadegesin R, Hinkes B, Saisawat P, Trevisson E, Doimo M, Casarin A, Pertegato V, Giorgi G, Prokisch H, Rotig A, Nurnberg G, Becker C, Wang S, Ozaltin F, Topaloglu R, Bakkaloglu A, Bakkaloglu SA, Muller D, Beissert A, Mir S, Berdeli A, Varpizen S, Zenker M, Matejas V, Santos-Ocana C, Navas P, Kusakabe T, Kispert A, Akman S, Soliman NA, Krick S, Mundel P, Reiser J, Nurnberg P, Clarke CF, Wiggins RC, Faul C, Hildebrandt F. COQ6 mutations in human patients produce nephrotic syndrome with sensorineural deafness. J Clin Invest. 2011 May;121(5):2013-24. doi: 10.1172/JCI45693. Epub 2011 Apr 11. PMID 21540551
- [Background] Alehagen U, Aaseth J, Larsson A, Alexander J. Decreased Concentration of Fibroblast Growth Factor 23 (FGF-23) as a Result of Supplementation with Selenium and Coenzyme Q10 in an Elderly Swedish Population: A Sub-Analysis. Cells. 2022 Feb 1;11(3):509. doi: 10.3390/cells11030509. PMID 35159318